CLINICAL TRIAL: NCT04451408
Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3372993 in Participants With Alzheimer's Disease and Healthy Participants
Brief Title: A Study of LY3372993 in Participants With Alzheimer's Disease (AD) and Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 17755; J1G-MC-LAKB (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease; Healthy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY3372993 (Part A) (Experimental): LY3372993 administered as multiple doses either intravenously (IV) or subcutaneously (SC).
  Interventions: Drug: LY3372993
- LY3372993 (Part B) (Experimental): LY3372993 administered as single dose IV or SC.
  Interventions: Drug: LY3372993
- Placebo (Part A) (Placebo Comparator): Placebo administered as multiple doses IV or SC.
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Placebo administered as single dose IV or SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3372993 — Administered IV or SC.
  Arms: LY3372993 (Part A); LY3372993 (Part B)
Drug: Placebo — Administered IV or SC.
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3372993 in participants with AD, non-Japanese, and Japanese healthy participants who are of first-generation Japanese origin. The study will also investigate how much LY3372993 gets into the bloodstream and will test the effects of LY3372993. The study will be conducted in two parts. The part A includes participants with AD and part B includes healthy participants. Participation could last up to about 61 weeks and may include up to 31 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

(Part A)

* Gradual and progressive changes in memory function reported by participants or their partners for greater than or equal to (≥) 6 months at screening, and a clinical diagnosis of mild cognitive impairment due to AD, or AD dementia, as determined by the investigator or based upon medical history
* Mini-Mental State Examination score ≥16
* Have clinical laboratory test results within normal reference range or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Have a study partner who will provide written informed consent to participate, is in frequent contact with the participant (defined as at least 10 hours per week), and will accompany the participant to study visits or be available through telephone at designated times

(Part B)

* overtly healthy males or females
* have a body mass index of 18.0 to 32.0 kg/m2, inclusive
* To qualify as a participant of the first-generation Japanese origin, the participant, the participant's biological parents, and all of the participant's biological grandparents must be of exclusive Japanese descent and born in Japan.

Exclusion Criteria:

(Part A)

* Have history or presence of uncontrolled asthma, significant autoimmune disease, hereditary angioedema, or known history of common variable immune deficiency
* Contraindication to positron emission tomography (PET)
* Have a history or presence of serious or unstable illnesses including cardiovascular, hepatic, renal, gastrointestinal, respiratory, endocrine, psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the analyses in this study, or increase risk for study intervention administration, or result in a participant's life expectancy of less than (<)24 months
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Have had significant medical history of dizziness, syncope, or vasovagal attacks within the past 3 years
* Contraindication to magnetic resonance imaging (MRI), including claustrophobia that cannot be managed with low-dose sedatives or the presence of contraindicated metal (ferromagnetic) implants/cardiac pacemaker

(Part B)

* have a family history of early onset AD (AD diagnosed prior to 65 years of age)
* have used or intend to use over-the-counter or prescription medication including herbal medications within 14 days prior to dosing.
* have a history or presence of significant psychiatric disorders
* have an abnormal blood pressure and/or pulse rate as determined by the investigator, or a pre-existing history of hypertension
* any clinically significant ECG or brain MRI abnormalities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Week 61 (part A) and Week 13 (Part B)
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3372993 | Day 1 Predose through Week 61 (part A) and Week 13 (Part B)
  PK: Cmax of LY3372993
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3372993 | Day 1 Predose through Week 61 (part A) and Week 13 (Part B)
  PK: AUC of LY3372993
Pharmacodynamics (PD): Change from Baseline in Cerebral Amyloid Plaque Level (Part A only) | Baseline and Week 61 (part A)
  PD: Cerebral amyloid plaque level measured using florbetapir positron emission tomography

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- United States (10):
  - Altasciences Clinical Los Angeles, Inc, Cypress, California
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Accel Research Sites- Clinical Research Unit, DeLand, Florida
  - MD Clinical, Hallandale, Florida
  - IMIC, Inc., Miami, Florida
  - Ppd Development, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Charter Research, The Villages, Florida
  - Synexus Clinical Research US, Inc., The Villages, Florida
  - Covance Dallas, Dallas, Texas
- Japan (3):
  - Oita University Hospital, Yufu, Oita Prefecture
  - The University of Tokyo Hospital, Bunkyo-ku, Tokyo
  - Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3372993 in Participants With Alzheimer's Disease (AD) — https://trials.lillytrialguide.com/en-US/trial/3qQDrJd2dTslGhNmqMga6Q